CLINICAL TRIAL: NCT06354959
Title: Prehab for Lung and Esophageal Cancer: Optimizing Well-being for Better Outcomes
Brief Title: Prehab for Lung and Esophageal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1030020
Record Dates: First submitted 2024-02-21; First posted 2024-04-09 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Neoplasm of Lung; Neoplasms; Exercise; Surgery
MeSH Terms: conditions — Lung Neoplasms; Neoplasms; Motor Activity | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Receive standard of care
- Prehab (Experimental): Complete an 8-week community based prehab program.
  Interventions: Behavioral: Prehabilitation

INTERVENTIONS:
Behavioral: Prehabilitation — 8-week community based prehab program
  Arms: Prehab

SUMMARY:
Research indicates that individuals diagnosed with lung or esophageal cancer who enter treatment with higher functional capacities, improved body composition, and better nutrition status tend to experience better outcomes and a higher quality of life. The primary objective of a prehabilitation health coaching program is to enhance the overall health and well-being of patients before they undergo major surgery.This personalized 8-week program encompasses elements such as nutrition, smoking cessation, sleep hygiene, and movement, equipping participants with the knowledge and tools needed to adopt healthier lifestyles.

DETAILED DESCRIPTION:
The purpose of this study is to explore the implementation, feasibility and effectiveness of a community-based prehabilitation health coaching program, including nutrition, smoking cessation, sleep hygiene and movement for individuals scheduled to undergo surgery for lung or esophageal cancer.. Participants will have the option to engage in a one-on-one prehabilitation health coaching program tailored to their needs, led by a Qualified Exercise Professional (QEP). The personalized prehabilitation plan will encompass 4-6 in-person or virtual meetings before surgery, including a structured movement plan, education on smoking cessation, sleep quality, stress reduction, mindfulness, and nutrition. Post-surgery, the QEP will provide support through counselling and scheduled sessions for a month after surgery and include one session while the patient is in hospital.

This research adopts a repeated measure, mixed-methods approach. Participants will undergo three clinical assessments at different stages: baseline, pre-surgery, and 4-6 weeks post-surgery. The findings from this study will guide future grant applications aimed at funding larger studies and the implementation of prehabilitation as part of standard of care in lung and esophageal cancer patients in Nova Scotia.

Central to the research endeavor is the driving question: "How can a community-based prehabilitation program be successfully implemented in the community, and can it lead to improved functional outcomes in patients undergoing surgery for lung or esophageal cancer?" This overarching question provides the study with its core focus and serves as a guiding force throughout the research process.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with lung or esophageal cancer
* Scheduled to receive surgical intervention in minimum 2-weeks
* Surgeon approval
* Able to read and write in English
* >18 years of age

Exclusion Criteria:

* Not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility- Recruitment | 2 years
  Participant accrual as defined as the number of eligible participants who consent to participate
Feasibility- Participant fidelity | 2 years
  Participant adherence to prescribed exercise intervention
Feasibility - Safety | 2 years
  Adverse and serious adverse events
Feasibility - Retention/Attrition | 2 years
  Percentage of participants who complete the 12-week intervention
Feasibility - Participant Experience | 2 years
  Exit interview is used to assess factors influencing participant selection of intervention type/setting, adherence to and satisfaction with the health coaching program
Feasibility- Attendance | 2 years
  Attendance is calculated as the percentage of exercise sessions completed by the total number of available exercise sessions over the 8-10-week intervention.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - Lung OR Esophageal (FACT-L/ FACT- E) | 8-10 week change
  44 item that measures multidimensional quality of life
Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | 8-10 week change
  a 13-item questionnaire that evaluates an individual's self-reported fatigue during their usual daily activities over the past week
5x chair stand | 8-10 week change
  To test functional strengths, risk of falling and overall leg strength and endurance
Stair climb test | 8-10 week change
  To test functional strength, balance and agility
Grip strength | 8-10 week change
  To test overall body strength
Resting Heart rate | 8-10 week change
  Resting heart rate
Resting blood pressure | 8-10 week change
  resting systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria General Hospital, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Langley JE, Sibley D, Chiekwe J, Keats MR, Snow S, Purcell J, Sollows S, Hill L, Watton D, Gaudry AE, Hashish I, Wallace A. Prehabilitation Program for Lung and Esophageal Cancers (Boosting Recovery and Activity Through Early Wellness): Protocol for a Nonrandomized Trial. JMIR Res Protoc. 2025 Mar 10;14:e60791. doi: 10.2196/60791. PMID 40063931